CLINICAL TRIAL: NCT00989417
Title: Effectiveness and Cost Of ICD Follow-up Schedule With Telecardiology
Brief Title: Benefits of Implantable Cardioverter Defibrillator Follow-up Using Remote Monitoring
Acronym: ECOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sophie FAUQUEMBERGUE, BIOTRONIK France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FRA041
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Implantable Cardioverter-Defibrillators; Ventricular Fibrillation; Tachycardia, Ventricular
Keywords: Remote monitoring; Defibrillators, Implantable; Home monitoring; Shock; Implantable cardioverter-defibrillator Therapy
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular; Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CONTROL Group - Without Home Monitoring (Active Comparator): Patients receiving the standard of care. Due to safety concerns, the patients are followed every 6 months after a first follow-up, which is performed between 1 and 3 months after implantation.
  Interventions: Other: ACTIVATION of HOME MONITORING
- ACTIVE GROUP With Home Monitoring (Experimental): After a first follow-up (between 1 and 3 months after implantation), the patients are followed one time per year. Within this period, the additional ICD follow-up or therapeutic intervention will be primarily triggered on cardio-reports reception, Data/IEGM-online analysis on internet site or patient/physician call.
  Interventions: Other: ACTIVATION of HOME MONITORING

INTERVENTIONS:
Other: ACTIVATION of HOME MONITORING — Both patient groups will be followed for 27 months and will have Home Monitoring switched on. The data from the CONTROL group will not be presented online to the attending physician, but a retrospective analysis on differences between the two groups will be performed.

SUMMARY:
In many aspects of every-day life, modern communication systems bring about a remarkable increase in comfort and safety by transmitting data and information in an easy and reliable manner. In order to provide these advantages also to patients with implantable cardioverter-defibrillators, as well as to their physicians, BIOTRONIK has developed a long-distance implant telemetry to enable periodic trend and event-triggered transmissions of implant data and intracardiac electrogram over distances of several meters. The data is received by a patient device and subsequently automatically transferred to a BIOTRONIK Service Center that provides it to the physician on a password secured internet site. Hence, the physician receives diagnostic information without the patient having to visit the physician (Home Monitoring, HM). New possibilities will arise for a detailed medical and event-correlated supervision of the patient's therapy using electrically active implants.

DETAILED DESCRIPTION:
State-of-the-art implantable cardioverter defibrillators (ICD) provide a variety of algorithms to optimize episode classification and to minimize the danger of delivering inadequate therapies. An important role in checking the correctness of episode detection, classification and treatment plays the intracardiac electrogram (IEGM), which is stored inside the ICD for every detected episode. However, to analyze the stored IEGM, the physician has to interrogate the implant, i.e. the patient has to visit the ICD ambulance for follow-up. As a result, follow-ups are performed principally to corroborate that the ICD has correctly classified and treated detected tachycardia episodes, to optimize the parameters and in case of adverse event detection, to modify the programmation.

The extension of BIOTRONIK Home Monitoring® by IEGM-Online® with LUMOS ICD offers a new possibility to meet the following challenge:

Due to its integrated long-distance telemetry, the implantable cardioverter defibrillator (ICD) LUMOS is capable of periodically transmitting data and IEGM-online from the ICD memory to the BIOTRONIK Service Center via patient device. The BIOTRONIK Service Center decodes the data and presents it to the physician on a password secured internet site. Additionally, in case certain event criteria are met, the most important Home Monitoring information is immediately faxed to the physician as an Event Report. These events can be customized by the physician. Thus, the physician will be able to closely monitor the patient and check the adequacy and efficiency of the ICD therapy without requiring the patient to visit the physician. The transmitted data comprise information on atrial and ventricular rhythm, atrioventricular conduction and system status.

The purpose of the present study is to evaluate the safety and economic impact of ICD follow-up schedule with Home Monitoring in France. For this assessment, the investigation compares two groups: For the ACTIVE group, after a first follow-up, the patients are only followed by Home Monitoring and one follow-up per year. The ICD follow-up or therapeutic intervention will be primarily based and triggered on event reports reception and after cardio reports and IEGM-online analysis on internet site. The findings from this group will be compared to those of a group receiving standard of care (CONTROL group). Both patient groups will be followed for 27 months and will have Home Monitoring switched on. The data from the CONTROL group will not be presented online to the attending physician, but a retrospective analysis on differences between the two groups will be performed. The clinical study will analyse, the incidence of significant serious adverse events (composite of all-cause mortality, cardiac and device related SAE), the costs reduction, the home-monitoring workload, the quality of life, the incremental Costs/Effectiveness ratio, the patient willing-to-pay, the delay of Home Monitoring to manage adverse events, the sensitivity of Home Monitoring to detect ICD dysfunctions, the inappropriate therapies rate and impact on hospitalization, the number of ICD charge and impact on battery longevity.

The trial will be conducted as a prospective, randomized, open, multicenter, national clinical trial. The enrolment of 400 patients in 40 clinical centres in France is anticipated

ELIGIBILITY:
Inclusion Criteria:

* Indication for single or dual chamber ICD

Exclusion Criteria:

* NYHA class IV
* Pregnant woman or woman who plan to become pregnant during the trial
* Patient whose medical situation is not stable
* Presence of any disease, other than patient's cardiac disease, associated with reduced likelihood of survival for the duration of the trial, e.g. cancer, uraemia (urea > 70mg/dl or creatinine >3mg/dl), liver failure, etc.
* Age < 18 years
* Patient unable to handle Home Monitoring system correctly
* The patient is not willing and able to comply with the protocol
* Change of residence expected during study
* Insufficient GSM coverage at patient's home
* Participation in another clinical study
* Patient unwilling to sign the consent for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2007-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with more than one Significant Serious Adverse Event (SSAE) since home-monitoring activation. SSAE is a composite comprising all-cause mortality, cardiac or device related Serious Adverse Events | 27 months

SECONDARY OUTCOMES:
Total costs minimization analyse | 27 months
Delay of Home Monitoring to manage adverse events | 27 months
Sensitivity of Home Monitoring to detect ICD dysfunction | 27 months
Number of capacitor charge and incidence on ICD-battery longevity | 27 months
Difference of cardiac and device related Adverse Event | 27 Months

CONTACTS AND LOCATIONS:
Overall Officials: Salem S KACET, Prof. Dr., Principal Investigator — CHRU de Lille- Hôpital Cardiologique - F 59037Lille -FRANCE
Locations (1):
- CHRU de Lille- Hôpital Cardiologique, Lille, France

REFERENCES:
- [Derived] Guedon-Moreau L, Lacroix D, Sadoul N, Clementy J, Kouakam C, Hermida JS, Aliot E, Kacet S; ECOST trial Investigators. Costs of remote monitoring vs. ambulatory follow-ups of implanted cardioverter defibrillators in the randomized ECOST study. Europace. 2014 Aug;16(8):1181-8. doi: 10.1093/europace/euu012. Epub 2014 Mar 9. PMID 24614572
- [Derived] Guedon-Moreau L, Kouakam C, Klug D, Marquie C, Brigadeau F, Boule S, Blangy H, Lacroix D, Clementy J, Sadoul N, Kacet S. Decreased delivery of inappropriate shocks achieved by remote monitoring of ICD: a substudy of the ECOST trial. J Cardiovasc Electrophysiol. 2014 Jul;25(7):763-70. doi: 10.1111/jce.12405. Epub 2014 Apr 10. PMID 24602062
- [Derived] Guedon-Moreau L, Lacroix D, Sadoul N, Clementy J, Kouakam C, Hermida JS, Aliot E, Boursier M, Bizeau O, Kacet S; ECOST trial Investigators. A randomized study of remote follow-up of implantable cardioverter defibrillators: safety and efficacy report of the ECOST trial. Eur Heart J. 2013 Feb;34(8):605-14. doi: 10.1093/eurheartj/ehs425. Epub 2012 Dec 13. PMID 23242192